CLINICAL TRIAL: NCT03537209
Title: Assessment of Root Apex Position of Mandibular Molars and Premolars Linear to Inferior Alveolar Canal Among a Sample of Egyptian Population Using CBCT: A Cross Sectional Study
Brief Title: Assessment Root Apex Position of Mandibular Molars and Premolars Linear to Inferior Alveolar Canal Among Egyptian Population Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Farid Medhat, Assistant Professor of Oral & Maxillofacial Radiology, Faculty of Dentistry, Cairo University
Other Study IDs: Rad 2:5:1
Record Dates: First submitted 2018-05-10; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Linear Measurement Between Roots of Mandibular Premolars & Molar & IAC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Linear relation between premolars and molars root apex and superior border of inferior alveolar canal

DETAILED DESCRIPTION:
The aim of the study is to assess the linear position between the roots of mandibular premolars and molars and the superior border of inferior alveolar canal.

Population: Adults, male and female from Egyptian population Outcome Variable: Linear measurement of the distance between root apices of mandibular premolars and molars to the superior border of IAN.

Outcome Measured Measuring Device Measuring Unit

Primary Outcome Distance between root apices of mandibular premolars and molars to inferior alveolar canal CBCT software Romexis® Millimeters

Research question:

Among the mandibular premolars and molars, which roots are the closest to the inferior alveolar canal, in sample of Egyptian Population?

Materials and Methods

Study Design: Cross-sectional Study

Setting and Location:

1. The data collection will be obtained from the data base available at Oral & Maxillofacial Radiology department at faculty of Dentistry, Cairo University.
2. CBCT images will be obtained from Egyptian patients who had CBCT examination as part of their dental examination, diagnosis or treatment planning during the years 2018.

Participants:

A total of 162 CBCT scans of mandibular permanent premolars and molars belonging to Egyptian individuals are selected according to the following:

Inclusion criteria:

* First and second mandibular permanent premolars and molars of Egyptian patients starting from 18 years, males or females.
* Intact roots without fractures or cracks.
* Posterior teeth are present and their adjacent and opposing teeth.
* Absence of radiological evidence of dental malocclusion that could have altered the position of premolars or molars.
* CBCT scans of mandibular first and second premolars and molars using 20 x 10 cm FOV, 0.4mm voxel resolution.

Exclusion criteria:

* Evidence of apicectomy or periapical surgery.
* Odontogenic or non-odontogenic pathology.
* Congenital deformity of the mandible.
* External Root resorption.
* Previous history of fracture of the mandible.
* Tomographic images of poor quality or artifacts interfering with the detection of mandibular canal and apical morphology of the teeth.

Variables:

1. The crowding and overlapping of the mandibular posterior teeth .
2. Extraction of the adjacent or the opposing tooth may cause tilting of the tooth or over eruption of the opposing tooth.
3. Attrition of the teeth may cause over eruption of the teeth.
4. The presence of dental anamolies may influence the position of the tooth to the inferior alveolar canal.

Data Sources / Measurements:

Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database by convenient sampling technique.

CBCT images will be obtained from patients who required CBCT examination as part of their dental examination, diagnosis or treatment planning without exposing them to unnecessary radiation dose for the research purpose.

All the CBCT examinations are scanned by Planmeca Promax 3D®, 20 x 10 cm FOV, 0.4 mm voxel resolution, 90 kVp, 8 mA and 13.5 seconds exposure time.

To assess the shortest distance from the root apices to the border of the inferior alveolar canal, the multiplanar reconstruction view of the manufacturer's software viewer (Planmeca Romexis) with its axial, sagittal and coronal plane will be used, and the cross-sectional images through the mandible will be also used.

Cross sectional images will be oriented parallel to the long axis of the tooth, then the shortest distance from the deepest point of root apices and superior border of the inferior alveolar canal will be obtained to be examined (Umut et al 2017).

CBCT images will be interpreted by two oral radiologists independently; blinded from demographic data of the patients and from the results of each other.

All measurements will be assessed, once by the first investigator and then another time two weeks later for intra-observer reliability. The second investigator will assess the measurements once for inter-observer reliability.

Then inter-observational and intra-observational variability between the observers will be evaluated.

Bias:

No source of bias.

Study Size:

The aim of the study is to assess the relationship between the roots of mandibular premolars and molars and the superior border of inferior alveolar canal in Egyptian population. Based on the previous paper by San Chong,et al,2017,the prevalence of alveolar nerve 78%.Using a precision of 5, a design effect set at 1 with 95%CI(confidence interval), a total sample size of 162 will be sufficient. The sample size was calculated by Epi info.

Sampling Strategy: The sample will be collected by convenient sampling technique.

Statistical Methods:

Data will be analyzed using IBM SPSS advanced statistics ( Statisitcal Package for Social Sciences), version 24 (SPSS Inc.,Chicago,IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percantages. Comparsions between male and females for normally distributed numeric variables will be done using Student's t-test while for non-normally distributed numeric variables will be done by Mann-Whitney test. Comparisons between categorical variables will be performed using the chi square test, A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be tailed.

ELIGIBILITY:
Inclusion Criteria:

* First and second mandibular permanent premolars and molars of Egyptian patients starting from 18 years, males or females.
* Intact roots without fractures or cracks.
* Posterior teeth are present and their adjacent and opposing teeth.
* Absence of radiological evidence of dental malocclusion that could have altered the position of premolars or molars.
* CBCT scans of mandibular first and second premolars and molars using 20 x 10 cm FOV, 0.4mm voxel resolution.

Exclusion Criteria:

* Evidence of apicectomy or periapical surgery.
* Odontogenic or non-odontogenic pathology.
* Congenital deformity of the mandible.
* External Root resorption.
* Previous history of fracture of the mandible.
* Tomographic images of poor quality or artifacts interfering with the detection of mandibular canal and apical morphology of the teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian population
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Distance between root apices of mandibular premolars and molars to inferior alveolar canal | 2018
  measurement in millimeters using CBCT software Romexis®

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03537209/Prot_000.pdf